CLINICAL TRIAL: NCT03307642
Title: Evaluation of a Text Based Reminder Recall System to Increase Utilization of the School Kids Influenza Prevention Project and Increase Influenza Vaccination Rates in Monroe County, NY
Brief Title: Evaluation of the School Kids Influenza Prevention Project
Acronym: SKIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Stanley J Schaffer, MD, Primary Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Version 3.01
Record Dates: First submitted 2017-10-05; First posted 2017-10-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Childhood Influenza Vaccination; School-located Influenza Vaccination
Keywords: Influenza vaccination rates; Respiratory Tract Diseases
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: SLIV will be offered at all schools in an urban school district. Students will be randomized into either SLIV + standard communication about SLIV or SLIV + standard communication + text message reminders.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLIV + usual communication (No Intervention): Parents receive usual communication from school (paper consent packets & automated voice mails) about SLIV
- SLIV + usual communication + text (Active Comparator): Parents receive usual communication from school (paper consent packets & automated voice mails) about SLIV plus a series of text messages informing them about the usual communication for SLIV
  Interventions: Other: Text message notification

INTERVENTIONS:
Other: Text message notification — Three text messages will be sent to 50% of the parents, scheduled around the standard methods of communication
  Arms: SLIV + usual communication + text

SUMMARY:
Children whose parents receive text reminders are more likely to be consented to participate in the school located influenza vaccination clinic than children whose parents do not receive text reminders.

ELIGIBILITY:
Inclusion Criteria:

- Enrolled in the urban school district

Exclusion Criteria:

- Attends a school in the urban district containing a school-based health center

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18540 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination status | Through January, 2018
  Vaccination status for the 2017/2018 influenza season will be assessed. The vaccination date will be recorded, as well as the provider name, to determine whether vaccine was received at the school-located influenza clinic

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Schaffer, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No